CLINICAL TRIAL: NCT00463710
Title: Effect of Interferon Beta-1a (Avonex®) on Changes of Non-conventional MRI Measures in Patients With Relapsing-remitting and Secondary-progressive Multiple Sclerosis
Brief Title: Effect of Interferon Beta-1a (Avonex®) on Changes of Non-conventional MRI Measures in Patients With MS
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Bianca Weinstock-Guttman, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 003-05-AVX
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
Keywords: MTI, DWI, Avonex, MRI
MeSH Terms: conditions — Multiple Sclerosis; Driving Under the Influence

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avonex® monotherapy (6.0 MIU administered i.m. each week)

SUMMARY:
Phase IV open label, single-blind study, post-marketing, 1-year MRI observational study evaluating effect of Avonex® monotherapy (6.0 MIU administered i.m. each week) on the year-to-year changes in two annual measures-magnetization transfer imaging and diffusion-weighted imaging in patients with either relapsing-remitting (RR) or secondary-progressive (SP) multiple sclerosis (MS). One hundred fifty (150) patients with RR and SP MS-followed at the Jacobs Neurological Institute, University at Buffalo, Buffalo NY-who satisfy both inclusion and exclusion criteria will be included. They will be assessed at baseline and at 12 months with MRI and clinical examinations.

DETAILED DESCRIPTION:
1.1. Protocol Title: Effect of Interferon beta-1a (Avonex®) on changes of non-conventional MRI measures in patients with relapsing-remitting and secondary-progressive multiple sclerosis.

1.2. Study rationale: Only a few longitudinal studies have investigated the effect of disease-modifying (DMT) on annual changes of non-conventional magnetic resonance imaging (MRI) measures, such as magnetization transfer imaging (MTI) in patients with multiple sclerosis (MS). In a previous study, the effect of interferon beta-1a (Avonex®) administered IM each week was investigated on the evolution of monthly magnetization transfer ratio (MTR) within new gadolinium (Gd)-enhancing lesions in patients with very early relapsing-remitting (RR) MS. Eight untreated patients with RRMS who completed up to 14 monthly brain MRI sessions elected to initiate treatment with Avonex®. The difference between MTR at appearance of 47 new Gd+ lesions before treatment versus 23 new Gd+ lesions during treatment with Avonex® was not significant. However, after appearance of new Gd+ lesions, the rate of increase in MTR (index of remyelination) was faster during therapy (p = 0.037). This study indicated that MTR abnormalities within new Gd+ lesions may evolve at a slower rate during treatment with Avonex® than before initiating therapy and that Avonex® may promote resolution of new Gd+ lesions. However, although this study yielded some positive results, it was not empowered to establish whether Avonex® may have a real treatment effect on lesion recovery. Moreover, in that study, the effect of Avonex® was not investigated on changes in normal appearing brain tissue (NABT) over time.

1.3. Study Aims: Aim 1. To define the effect of interferon beta-1 (Avonex®) monotherapy (6.0 MIU administered i.m. each week) on the year-to-year changes in two annual measures-MTI and diffusion-weighted imaging (DWI)-in patients with either RR or secondary-progressive (SP) MS.

Aim 2. To explore differences in the progression of these two non-conventional MRI measures between patients who do and do not develop significant brain atrophy, hyperintense T2- and hypointense T1 (black holes) lesion volume (LV) progression during the same 12 months.

Aim 3. To investigate differences in the progression of non-conventional MRI measures between patients who respond or not respond to Avonex® monotherapy during the same 12 months.

1.4. Design and Methods: 1.4.1. Study outline: Phase IV open label, single-blind study, post-marketing, 1-year MRI observational study evaluating effect of Avonex® monotherapy (6.0 MIU administered i.m. each week) on the year-to-year changes in two annual measures-MTI and DWI-in patients with either RR or SP MS.

One hundred fifty (150) patients with RR and SP MS-followed at the Jacobs Neurological Institute, University at Buffalo, Buffalo NY-who satisfy both inclusion and exclusion criteria will be treated with Avonex® monotherapy. They will be assessed at baseline and at 12 months with MRI and clinical examinations. These patients are part of a larger cohort of MS patients (1000) who are on Avonex® mono- or combination therapy and are being routinely followed at the Jacobs Neurological Institute.

MRI assessment will include detailed conventional and non-conventional protocol. Neurological assessment included Kurtzke Expanded Disability Status Scale (EDSS) score and evaluation of relapses.

1.4.2. Outcome measures: The primary outcome of the study is to measure the effect of Avonex® monotherapy on changes in lesional MTR, whole brain (WB) MTR, normal appearing GM (NAGM) MTR and normal appearing WM (NAWM) MTR, as well as in WB mean diffusivity (MD) and entropy, as measured by the 1-year changes from baseline.

The secondary outcomes will include measurement of brain parenchymal fraction (BPF), GM fraction (GMF), WM fraction (WMF), T1- and T2- (LV), number and volume of Gd-enhancing lesions and evaluation of annual relapse rate and EDSS.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with clinical definite MS according to the McDonald criteria
* Age 18-65
* Have a RR or SP disease course
* Have EDSS scores less than or equal to 6.5
* Have disease duration 6 months to 20 years
* Be on intramuscular 6 MIU of Avonex® for a minimum of 3-6 months before the study entry
* Signed informed consent
* None of the exclusion criteria

Exclusion Criteria:

* Previous treatment 3 months prior to study entry with immunosuppressant agents, e.g., mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine or total body irradiation or any other concomitant immunomodulatory therapies besides Avonex® (e.g., Azathioprine, methotrexate, IVIG, cellcept, natalizumab, etc).
* Patients who received steroid therapy during the 3 months prior to study entry or patients who received steroid treatment 30-60 days prior to the follow-up MRI scan date.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-06; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — SUNY Buffalo
Locations (1):
- The Jacobs Neurological Institute, Buffalo, New York, United States